CLINICAL TRIAL: NCT02199704
Title: Self Directed Positive Parenting Program (Triple P) for Psychosis: A Clinical Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Lancashire Care NHS Foundation Trust (Network)
Responsible Party: Principal Investigator, Dr Chris Taylor, Clinical Psychologist, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 14/NW/0126
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2015-11

CONDITIONS: Schizophrenia; Spectrum; Disorders
Keywords: Parenting; Psychosis; Schizophrenia; Delusions; Hallucinations
MeSH Terms: conditions — Schizophrenia; Disease; Psychotic Disorders; Delusions; Hallucinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No control or comparison arm. (Other): This case series study has no control or comparison arm. There is only one arm being evaluated (the self directed parenting intervention).
  Interventions: Other: Self Directed Positive Parenting Program

INTERVENTIONS:
Other: Self Directed Positive Parenting Program — Individuals with psychosis who are parents will receive a copy of the "Every Parent's Self Help Workbook" (Markie-Dadds, Sanders & Turner, 1999) and up to ten sessions of support. This is a case series study.
  Other Names: "Every Parent's Self Help Workbook"

SUMMARY:
The aim of the case series study is to explore if a self directed version of the Positive Parenting Program (Triple P) is a feasible and acceptable intervention for individuals with psychosis who are parents.

DETAILED DESCRIPTION:
As above.

ELIGIBILITY:
Inclusion Criteria:

* 1. Parents/caregivers (mothers or fathers) with a Schizophrenia-spectrum diagnosis who are:

  2. Aged 18 years or more

  3. Have at least one child aged 3-10 years old

  4. Have a least 10 hours contact time per week with the child.

  5. Identify difficulties in parenting during assessment

Exclusion Criteria:

* 1. Parents/caregivers and family members who do not have good working knowledge of English. They should have enough practical experience to be able to adequately use the English language to understand and respond to questions, to read and complete questionnaires

  2. Families who do not have at least one adult who has basic literacy skills

  3. Families where there is known intention for their children to be taken into care or where the parent(s) have no regular contact with the index child

  4. Parents with a clinical schizophrenia-spectrum diagnosis who have recently been discharged from acute in-patient care for their condition and have less than four weeks of stabilisation of psychotic experiences (operationally defined as no significant change to management or severity of symptoms in a four-week period since discharge as assessed from case notes). This is because if a potential parent with schizophrenia had recently required an inpatient stay, it is important to give them sufficient time to readjust to living in the community and ensure sufficient time is provided for symptom stabilisation before taking part

  5. Families seeking support from services regarding child management issues

  6. Families actively involved in another current cognitive behavioural therapy based intervention

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The Psychotic Symptom Rating Scales (PSYRATS) | Initial Ax, Multiple Baseline Ax, Final Baseline Ax, Up to 10 support sessions Ax, End Ax, Follow Up Ax. Ax from 0 - 16 weeks.
  Ax from 0 - 16 weeks.
Parenting and Family Adjustment Scale (PAFAS) | Initial Ax, Multiple Baselines, Final Baseline, Support Sessions, End Ax, Follow Up. Ax from 0 - 16 weeks.
  Ax from 0 - 16 weeks.

SECONDARY OUTCOMES:
Eyberg Child Behaviour Inventory (ECBI) | Initial Ax, Final Ax, End Ax, Follow Up. Ax from 0 - 16 weeks.
  Ax from 0 - 16 weeks.
Parenting Task Checklist (PTC) | Initial Ax, Final Ax, End Ax, Follow Up. Ax from 0 - 16 weeks.
  Ax from 0 - 16 weeks.
Depression Anxiety and Stress Scale (DASS-21) | Initial Ax, Final Ax, End Ax, Follow Up. Ax from 0 - 16 weeks.
  Ax from 0 - 16 weeks.
Work and Social Adjustment Scale (WSAS) | Initial Ax, Final Ax, End Ax, Follow Up. Ax from 0 - 16 weeks.
  Ax from 0 - 16 weeks.
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Initial Ax, Final Ax, End Ax, Follow Up. Ax from 0 - 16 weeks.
  Ax from 0 - 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Rachel Calam, PhD, Study Chair — University of Manchester
Locations (1):
- University of Manchester, Manchester, United Kingdom